CLINICAL TRIAL: NCT05110001
Title: Rose Bengal Electromagnetic Activation With Green Light for Infection Reduction
Acronym: REAGIR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Aravind Eye Care System (Other); National Eye Institute (NEI) (NIH); Stanford University (Other); Federal University of São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18-26045-R; UG1EY028518 (NIH)
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Results first posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Acanthamoeba Keratitis; Fungal Keratitis
MeSH Terms: conditions — Acanthamoeba Keratitis | interventions — chlorhexidine gluconate; Natamycin; Rose Bengal; Corneal Cross-Linking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Therapy (Placebo Comparator): Patients in this arm will receive topical chlorhexidine gluconate 0.02% (acanthamoeba), moxifloxacin 0.5% (smear/culture negative) or natamycin 5% (fungal keratitis) plus sham RB-PDT
  Interventions: Drug: Moxifloxacin Ophthalmic; Drug: Chlorhexidine Gluconate; Drug: Natamycin; Other: Placebo
- Cross-Linking with rose Bengal (RB-PDT) (Experimental): Patients in this arm will receive topical chlorhexidine gluconate 0.02% (acanthamoeba), moxifloxacin 0.5% (smear/culture negative) or natamycin 5% (fungal keratitis) plus RB-PDT
  Interventions: Drug: Moxifloxacin Ophthalmic; Drug: Chlorhexidine Gluconate; Drug: Natamycin; Drug: Rose Bengal

INTERVENTIONS:
Drug: Moxifloxacin Ophthalmic — Topical moxifloxacin 0.5% is a fluoroquinolone antibiotic that is used to treat bacterial infections. This is a standard therapy for bacterial keratitis.
Drug: Chlorhexidine Gluconate — Topical chlorhexidine gluconate 0.02% is an antiseptic agent, with both antibacterial and antifungal properties. This is a standard therapy for Acanthamoeba keratitis.
Drug: Natamycin — Natamycin 5% is an antifungal agent used to treat fungi that cause keratitis. This is a standard therapy for fungal keratitis.
Drug: Rose Bengal — Study participants receive RB-PDT within 48 hours of randomization. All participants will receive a 30-minute loading dose of topical Rose Bengal (0.1% RB in 0.9% sodium chloride) which will be applied in 5-minute intervals to the de-epithelialized cornea. This will be followed by irradiation with a 6mW/cm2 custom-made green LED source for 15 minutes (5.4J/cm2). Repeat cornea culture will be collected within 24 hours after the procedure.
  Other Names: Corneal Cross Linking with rose Bengal
  Arms: Cross-Linking with rose Bengal (RB-PDT)
Other: Placebo — Study participants receive sham RB-PDT within 48 hours of randomization. Participants will receive a 30-minute loading dose of topical balanced salt solution which will be applied in 5-minute intervals to the de-epithelialized cornea. A pen light covered with a green filter will be used for 15 minutes. Repeat cornea culture will be collected 30 minutes after the sham procedure.
  Arms: Standard Therapy

SUMMARY:
Rose Bengal Electromagnetic Activation with Green light for Infection Reduction (REAGIR ) is an international, randomized, doubled masked, clinical trial. The purpose of this study is to determine differences in 6-month visual acuity between medical antimicrobial treatments alone versus antimicrobial treatment plus cross-linking with rose Bengal (RB-PDT).

Patients presenting to one of the Aravind Eye Hospitals in India or to the Federal University of São Paulo ophthalmology clinic in Brazil with either smear or culture positive fungal or acanthamoeba keratitis or smear and culture negative corneal ulcers and moderate to severe vision loss, defined as Snellen visual acuity of 20/40 or worse, will be eligible for inclusion. Those who agree to participate will be randomized to one of two treatment groups:

Group 4, Sham RB-PDT: topical chlorhexidine gluconate 0.02% (acanthamoeba), moxifloxacin 0.5% (smear/culture negative) or natamycin 5% (fungal keratitis) plus sham RB-PDT

Group 5, RB-PDT: topical chlorhexidine gluconate 0.02% (acanthamoeba), moxifloxacin 0.5% (smear/culture negative) or natamycin 5% (fungal keratitis) plus RB-PDT.

ELIGIBILITY:
Inclusion Criteria:

* Presence of smear or culture positive fungal or acanthamoeba ulcer; smear or culture negative ulcer; or any atypical bacteria (such as Nocardia)
* Moderate to severe vision loss, defined as Snellen visual acuity of 20/40 (6/12) or worse
* Corneal thickness ≥350 µm, as measured on AS-OCT
* Age over 18 years
* Basic understanding of the study as determined by the physician
* Commitment to return for follow up visits

Exclusion Criteria:

* Evidence of concomitant infection on exam, gram stain, or confocal microscopy (i.e. herpes, both bacteria and acanthamoeba on gram stain)
* Impending or frank perforation at recruitment
* Involvement of sclera at presentation
* Non-infectious or autoimmune keratitis
* History of corneal transplantation
* History of intraocular surgery within last three months
* Pinhole visual acuity worse than 20/200 in the unaffected eye
* Participants who are decisionally and/or cognitively impaired
* Presence of demestocele at recruitment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2024-12-14 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lietman, MD, Principal Investigator — University of California, San Frnasco; Jennifer Rose-Nussbaumer, MD, Principal Investigator — Stanford University; Nicole Varnado, MPH, Study Director — Stanford University
Locations (2):
- Federal University of São Paulo, São Paulo, Brazil
- Aravind Eye Care System, Madurai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Christy SJ, Mandlik K, Kumar V, Kanchugantla SSSM, Abdelrahman S, Rose-Nussbaumer J. Adjunctive tacrolimus in the treatment of fungal keratitis requiring therapeutic penetrating keratoplasty. Am J Ophthalmol Case Rep. 2025 Dec 29;41:102506. doi: 10.1016/j.ajoc.2025.102506. eCollection 2026 Mar. PMID 41561665
- [Derived] Prajna NV, Lalitha P, Sharma S, de Freitas D, Hofling-Lima A, Varnado N, Abdelrahman S, Cavallino V, Arnold BF, Lietman TM, Rose-Nussbaumer J. A double-masked, sham-controlled trial of rose bengal photodynamic therapy for the treatment of fungal and acanthamoeba keratitis: Rose Bengal Electromagnetic Activation with Green Light for Infection Reduction (REAGIR) study. Trials. 2024 Aug 28;25(1):566. doi: 10.1186/s13063-024-08376-3. PMID 39192339
- [Derived] Prajna V, Prajna L, Sharma S, de Freitas D, Hofling-Lima AL, Varnado N, Abdelrahman S, Cavallino V, Arnold B, Lietman T, Rose-Nussbaumer J. A double-masked, sham-controlled trial of rose bengal photodynamic therapy for the treatment of fungal and acanthameoba keratitis: Rose Bengal Electromagnetic Activation with Green Light for Infection Reduction (REAGIR) Study. Res Sq [Preprint]. 2024 Jul 2:rs.3.rs-4165312. doi: 10.21203/rs.3.rs-4165312/v1. PMID 39011096

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Therapy | Cross-Linking With Rose Bengal (RB-PDT)
Started | 165 | 165
Completed | 149 | 148
Not Completed | 16 | 17

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Therapy | Cross-Linking With Rose Bengal (RB-PDT) | Total
Number analyzed (Participants) | 165 | 165 | 330
Number analyzed (Eyes) | 165 | 165 | 330
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (12) | 50 (13) | 50 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 59 | 117
  Male | 107 | 106 | 213
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 13
  Not Hispanic or Latino | 148 | 150 | 298
  Unknown or Not Reported | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 151 | 147 | 298
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 2 | 1 | 3
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 8 | 9 | 17
Visual Acuity (logMAR BSCVA) [Mean (Standard Deviation); unit: logMar] | 1.1 (0.50) | 1.2 (0.51) | 1.1 (0.50)
Central Corneal Thickness (μm) [Mean (Standard Deviation); unit: μm] | 630 (130) | 650 (130) | 640 (130)
Hypopyon [Count of Participants; unit: Participants]
  None | 99 | 87 | 186
  < 0.5 mm | 14 | 17 | 31
  Other | 52 | 61 | 113
Infiltrate/Scar Size (mm) [Mean (Standard Deviation); unit: mm] | 3.7 (1.4) | 3.8 (1.5) | 3.8 (1.4)
Fungal Culture (Positive) [Count of Participants; unit: Participants] | 118 | 115 | 233
Fungal Smear (Positive) [Count of Participants; unit: Participants] | 142 | 141 | 283
Acanthamoeba Culture [Count of Participants; unit: Participants]
  Positive | 6 | 2 | 8
  Negative | 54 | 54 | 108
  Not performed | 105 | 109 | 214
Acanthamoeba Smear (Postive) [Count of Participants; unit: Participants] | 4 | 1 | 5
Occupation [Count of Participants; unit: Participants]
  Manual Labor-Agriculture | 84 | 71 | 155
  Manual Labor- Non-Agriculture | 41 | 61 | 102
  Service/Clerical | 1 | 4 | 5
  Skilled Labor | 6 | 5 | 11
  Business/Trade | 3 | 1 | 4
  Domestic (Housework) | 7 | 2 | 9
  Student | 2 | 3 | 5
  Retired | 1 | 0 | 1
  Unemployed | 15 | 10 | 25
  Other | 5 | 8 | 13
Recent Eye Trauma [Count of Participants; unit: Participants] | 110 | 100 | 210
Contact Menswear [Count of Participants; unit: Participants] | 4 | 3 | 7
Uses Native Medicine [Count of Participants; unit: Participants] | 13 | 7 | 20
Symptom Duration (Days) [Mean (Standard Deviation); unit: days] | 8.0 (7.1) | 9.1 (8.9) | 8.5 (8.0)

OUTCOME MEASURES:

1. Primary Outcome: Best Spectacle-Corrected Visual Acuity
Description: Best Spectacle-Corrected Visual Acuity
Time Frame: 6 Months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Standard Therapy | Cross-Linking With Rose Bengal (RB-PDT)
Number analyzed (Participants) | 149 | 148
logMAR | 0.614 (0.658) | 0.666 (0.675)

2. Secondary Outcome: Best Spectacle-Corrected Visual Acuity
Description: Best Spectacle-Corrected Visual Acuity
Time Frame: 3 Weeks, 3 Months, 12 Months
Population: Loss to follow up
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Standard Therapy | Cross-Linking With Rose Bengal (RB-PDT)
Number analyzed (Participants) | 165 | 165
logMAR
  3-week: number analyzed (Participants) | 147 | 152
  3-week | 0.821 (0.630) | 0.855 (0.617)
  3-month: number analyzed (Participants) | 137 | 138
  3-month | 0.700 (0.661) | 0.772 (0.673)
  12- month: number analyzed (Participants) | 141 | 141
  12- month | 0.531 (0.662) | 0.611 (0.669)

3. Secondary Outcome: Scar Size
Description: Geometric Mean
Time Frame: 3 Weeks, 3 Months, 6 Months 12 Months
Population: Loss to follow up or CP/TPK
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Eyes
Arm/Group | Standard Therapy | Cross-Linking With Rose Bengal (RB-PDT)
Number analyzed (Participants) | 135 | 133
Number analyzed (Eyes) | 135 | 133
mm
  3-weeks | 3.84 (1.64) | 3.37 (1.35)
  3-months: number analyzed (Participants) | 126 | 120
  3-months: number analyzed (Eyes) | 126 | 120
  3-months | 3.99 (1.61) | 3.71 (1.52)
  6-months: number analyzed (Participants) | 135 | 128
  6-months: number analyzed (Eyes) | 135 | 128
  6-months | 3.96 (1.63) | 3.73 (1.53)
  12-months: number analyzed (Participants) | 128 | 128
  12-months: number analyzed (Eyes) | 128 | 128
  12-months | 3.65 (1.62) | 3.64 (1.43)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Standard Therapy | Cross-Linking With Rose Bengal (RB-PDT)
All-Cause Mortality (participants affected / at risk) | 1/165 | 0/165
Serious Adverse Events (participants affected / at risk) | 31/165 | 36/165
Other Adverse Events (participants affected / at risk) | 17/165 | 25/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy (N=165) | Cross-Linking With Rose Bengal (RB-PDT) (N=165)
Non-elective surgery, hospitalization, or loss of function (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic Penetrating Keratoplasty (Eye disorders) | 20 | 29
Corneal perforation (Eye disorders) | 2 | 2
Therapeutic Penetrating Keratoplasty and Corneal Perforation (Eye disorders) | 9 | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard Therapy (N=165) | Cross-Linking With Rose Bengal (RB-PDT) (N=165)
Increase in hypopyon (increase >2mm) (Eye disorders) | 6 | 7
Increase in the longest diameter of infiltrate (>50% increase from baseline and >1mm) (Eye disorders) | 10 | 14
Progressive corneal thinning, < 50% of enrollment thickness (Eye disorders) | 1 | 3
Other (Eye disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-09-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT05110001/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-03): https://cdn.clinicaltrials.gov/large-docs/01/NCT05110001/SAP_001.pdf